CLINICAL TRIAL: NCT01293942
Title: A Single-arm Phase II Downsizing Study of Irinotecan, Capecitabine and Oxaliplatin (IXO) and Bevacizumab as First-line Treatment to Assess Conversion to Resectability of Liver-only Metastases in Colorectal Cancer Patients With Initially Unresectable Metastases
Brief Title: IXO+A in mCRC With Liver-only Metastases
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Hoffmann-La Roche (Industry); Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OTT 10-01
Record Dates: First submitted 2011-02-08; First posted 2011-02-11 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Metastatic Colorectal Cancer
Keywords: unresectable liver-only metastases in colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Irinotecan; Capecitabine; Oxaliplatin; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IXO+A (Experimental): IXO regimen with Avastin
  Interventions: Drug: irinotecan, capecitabine, oxaliplatin (IXO) and bevacizumab

INTERVENTIONS:
Drug: irinotecan, capecitabine, oxaliplatin (IXO) and bevacizumab — IXO plus bevacizumab regimen is given every 3 weeks (Q3W), in the following order: Bevacizumab (A): 7.5 mg/kg via IV infusion, day 1 Oxaliplatin (O): 100 mg/m2 via 2-hour IV infusion, day 1 Irinotecan (I): 160 mg/m2 via 1-hour IV infusion, day 1 Capecitabine (X): 950 mg/m2 twice daily PO, days 2 - 15

SUMMARY:
The percentage of patients with defined unresectable metastatic disease who will benefit from a first-line treatment enabling secondary complete metastasectomy is unknown but limited. Definition of optimized treatment algorithms is difficult due to very inhomogeneous patient populations.

This open label, multicentre Phase II study primarily aims to assess the resection rate achievable in a selected patient population with initially unresectable metastatic disease limited to the liver only in order to evaluate feasibility, safety and efficacy with regards to secondary resection of hepatic lesions in these patients.

The trial aims to enrol only patients meeting defined criteria of unresectability with regards to their hepatic lesions and will exclude patients with extrahepatic lesions in order to examine the most appropriate, highly active treatment regimen for this group of unresectable patients with the highest probability of a successful secondary metastasectomy with curative intent. The trial will be conducted in highly specialized centres with a track record of successful interdisciplinary treatment approaches in the field of metastatic colorectal cancer to allow the precise assessment of the peri-operative safety parameters as well as an evaluation of the surgical treatment approaches.

The IXO regimen selected for this study has shown in a phase I/II study promising efficacy and a favourable safety profile. Bevacizumab has demonstrated a significant survival benefit in combination with chemotherapy in metastatic colorectal cancer. Therefore the study will allow evaluation of its potential benefit in combination with the two most active current chemotherapy regimens in the first-line and post-operative treatment setting.

ELIGIBILITY:
Inclusion Criteria:

* Primary colorectal cancer with unresectable metastatic lesion(s)
* At least one measurable lesion, confirmed by CT scan
* Male and female patients, aged ≥ 18 years
* ECOG performance score of 0 or 1 (within 1 week of study treatment start)
* Written informed consent
* Adequate general condition, cardiopulmonary functions and performance status
* Liver metastases no initially foreseen R0 resection of all hepatic lesions, but deemed potentially resectable after response to downsizing therapy

Exclusion Criteria:

* Extrahepatic metastatic disease
* Prior systemic or local treatment for metastatic disease, prior therapy with a biologic agent, prior adjuvant or neo-adjuvant chemotherapy, prior radiotherapy to the liver, other concurrent chemotherapy
* Inadequate bone marrow, liver, renal function, uncontrolled hypertension
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-03; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
conversion to resectability during downsizing therapy with IXO+A patients with initially unresectable liver-only metastases associated with colorectal cancer | after 8 IXO+A cycles

SECONDARY OUTCOMES:
Recurrence-free survival (RFS) | Every 2 cycles
Progression-free survival (PFS) | Every 2 cycles
Time to response (TTR) | Every 2 cycles
Overall survival (OS) | Every 2 cycles
Pathological complete response (pCR) rate | assessed post-operatory
Overall response rate (ORR) | Every 2 cycles
Number of participants with Adverse Events as a measure of Safety and Tolerability | Every 3 weeks
Surgical safety (frequency of surgical complications) | assessed post-operatory
Pathological changes in the non-tumoural liver following therapy with IXO+A | assessed post-operatory
R0, R1, R2 resection rate after up to 8 cycles of downsizing therapy with IXO+A | assessed post-operatory

CONTACTS AND LOCATIONS:
Overall Officials: Jean Maroun, MD, Study Chair — The Ottawa Hospital Cancer Centre
Locations (4):
- Canada (4):
  - The Ottawa Hospital Cancer Center, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec